CLINICAL TRIAL: NCT03850249
Title: Radioscapholunate Fusions After Wrist Trauma: Long-term Clinical and Radiographic Results.
Brief Title: Radioscapholunate Fusions After Wrist Trauma
Acronym: Radioscapho
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0010
Record Dates: First submitted 2019-01-24; First posted 2019-02-21 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Posttraumatic Radiocarpal Osteoarthritis
Keywords: Radioscapholunate; Fusion; Arthrodesis; Radiocarpal osteoarthritis; Partial radiocarpal fusion
MeSH Terms: conditions — Ankylosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators conduced a clinical trial to evaluate the clinical and radiographic results after radioscapholunate fusion in case of posttraumatic radiocarpal osteoarthritis.

Because of poor clinical result, many authors upgrade the procedure including excision of the distal pole of the scaphoid and later excision of the entire triquetrum.

Only one study compared the three procedures in 17 patients. The investigators performed the same comparison in 85 patients with a mean follow up of 9,1 years (1-23)

DETAILED DESCRIPTION:
The investigators compared three populations: patients with radioscapholunate (RSL) fusion alone, patients with RSLfusion and distal scaphoid excision and patient with RSL fusion, distal scaphoid excision and excision of the triquetrum.

The investigators performed clinical (pain, grasp strength, wrist motion), functional and radiographic (midcarpal osteoarthritis and radiocarpal nonunions) evaluation

ELIGIBILITY:
Inclusion criteria:

* posttraumatic radiocarpal osteoarthritis
* Patients who underwent radioscapholunate fusion

Exclusion criteria:

* Patients with radiocarpal osteoarthritis due to rheumatoid or inflammatory disease and Kienböck disease
* Patients with posttraumatic radiocarpal osteoarthritis managed with other surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had posttraumatic radiocarpal osteoarthritis and underwent RSL fusion
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
presence of mediocarpal osteoarthritis | 1 day
  To evaluate the long-term radiographic results of post-traumatic radio scapholunate
presence of scapho-trapezoidal trapezoid | 1 day
  To evaluate the long-term radiographic results of post-traumatic radio scapholunate
presence of non-consolidation of radio-scapho-lunar arthrodesis | 1 day
  To evaluate the long-term radiographic results of post-traumatic radio scapholunate

SECONDARY OUTCOMES:
Assess overall survival | 1 day
  To evaluate the overall survival (excluding total wrist arthrodesis) of post-traumatic radio scapholunate
the prognostic factors of good clinical | 1 day
  To evaluate the prognostic factors of good clinical (ie absence of osteoarthritis or good consolidation of arthrodesis)
the prognostic factors of radiographic evolution | 1 day
  To evaluate the prognostic factors of radiographic evolution (ie absence of osteoarthritis or good consolidation of arthrodesis)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Degeorge, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France